CLINICAL TRIAL: NCT03840187
Title: Correlation Between Colposcopist Findings and Digital Cervicography Employing Gynescope System
Status: Completed | Type: Observational
Sponsor: Barzilai Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 0097-18-BRZ
Record Dates: First submitted 2019-02-04; First posted 2019-02-15 (Actual); Last update posted 2020-01-18 (Actual); Status verified 2019-01

CONDITIONS: Cervical Dysplasia
Keywords: digital cervicography; Gynescope system
MeSH Terms: conditions — Uterine Cervical Dysplasia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Digital cervicography — Colposcopist findings and digital cervicography employing Gynescope system

SUMMARY:
Correlation between colposcopist findings and digital cervicography employing Gynescope system

DETAILED DESCRIPTION:
Up to 30 women that will be referred for colposcopy examination at the standard indications will also undergo a colposcopy examination of the cervix by a gynescope. The physicain performing the optical test will record the findings in accordance with the International Federation for Cervical Pathology and Colposcopy (IFCPC) terminology. Categorical variable will be included in every record. At later stage, the images obtained by the cervicography will be evaluated and recorded in accordance with the IFCPC terminology. Correlation between the categorical findings in both assesments will be compared. The correlation measure will be performed by Kappa test according to the categorial result of both measurements.

ELIGIBILITY:
Inclusion Criteria:

- Patients reffered for colposcopy

Exclusion Criteria:

Patient refusion

Ages: 18 Years to 65 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: Patients reffered for colposcopy
Sampling Method: Non-Probability Sample
Enrollment: 29 (Actual)
Dates: Start 2019-03-11 (Actual); Primary Completion 2020-01-15 (Actual); Study Completion 2020-01-15 (Actual)

PRIMARY OUTCOMES:
Categorical findings according in accordance with the International Federation of Cervical Pathology Colposcopy | 5 months
  leukoplakia, aceto - white change, mosaic, punctuation, and abnormal vessels

CONTACTS AND LOCATIONS:
Overall Officials: Ofer Gemer, Professor, Principal Investigator — Barzilai University Medical Center Ashkelon
Locations (1):
- Barzilay University Medical Center, Ashkelon, Israel